CLINICAL TRIAL: NCT00774891
Title: Comparison Of Left Ventricular Volume And Wall Stress With Dobutamine And Exercise Echocardiography
Status: Withdrawn | Type: Observational
Why Stopped: difficulty enrolling patients into this study
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-091
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Ischemia; Angina
Keywords: Echocardiography- exercise; Echocardiography- dobutamine; Wall stress; Ventricular volume-left; Ischemia; Angina; Heart diseases; Stress echocardiography; Ventricular volume; Vascular diseases
MeSH Terms: conditions — Ischemia; Angina Pectoris; Heart Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare the physiologic responses between exercise stress echocardiography and pharmacologic stress echocardiography on left ventricular volume and wall stress.

DETAILED DESCRIPTION:
This prospective observational study will compare the physiologic responses between exercise stress echocardiography and dobutamine stress echocardiography on left ventricular volume and wall stress. Exercise and dobutamine stress testing are two widely employed diagnostic modalities that are often used, interchangeably, to detect inducible ischemia. We hypothesize that dobutamine leads to significantly lower ventricular volumes and wall stress than exercise.

Some previous studies have shown that dobutamine and exercise echocardiography have comparable sensitivities and specificities, differences exist between the hemodynamic effects produced by each modality on the cardiovascular system. These variable effects may lead to differences in left ventricular size, volume and wall stress. If divergent left ventricular effects exist(between exercise and dobutamine induced stress), then the degree of myocardial oxygen consumption, ischemic burden, and ischemic threshold observed during exercise and dobutamine stress testing may be different between these commonly used modalities of stress testing.

The potentially variable effects on the left ventricle in response to the modality used to induce stress would highlight a physiological difference between exercise and dobutamine stress testing. Differences in volumes and stress could also help explain the greater of ischemia and higher frequency of angina and ST-segment deviation which has been previously observed in some studies during exercise as compared to dobutamine echocardiography. The presence or lack of these expected hemodynamic responses may also have additional diagnostic and prognostic implications.

The study involves the collection of data among patients undergoing stress echocardiograms that are clinically indicated. This data will be retrieved from the echocardiogram and report and medical chart, including baseline clinical characteristics, exercise parameters achieved during the test.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* Normal sinus rhythm on electrocardiogram
* Normal left ventricular systolic function on baseline echocardiogram

Exclusion Criteria:

* Patients with stress-induced wall motion abnormalities
* Left ventricular hypertrophy
* Evidence of prior myocardial infarction
* More than mild valvular heart disease
* Prior cardiac surgery
* Poor technical quality of echocardiogram

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lahey Clinic patients referred by their physician for stress echocardiograms for clinical indications. Approximately 30 patients referred for an exercise stress echocardiography and approximately 30 patients referred for a dobutamine stress echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Dobutamine stress echocardiography causes decrease in LV size/volume and wall stress compared to exercise stress echocardiography | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B. Labib, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Iwasaka T, Nakamura S, Sugiura T, Tarumi N, Yuasa F, Morita Y, Wakayama Y, Inada M. Difference between women and men in left ventricular pump function during predischarge exercise test after acute myocardial infarction. Am J Cardiol. 1994 Jan 1;73(1):11-5. doi: 10.1016/0002-9149(94)90719-6. PMID 8279370
- [Background] Mertes H, Erbel R, Nixdorff U, Mohr-Kahaly S, Kruger S, Meyer J. Exercise echocardiography for the evaluation of patients after nonsurgical coronary artery revascularization. J Am Coll Cardiol. 1993 Apr;21(5):1087-93. doi: 10.1016/0735-1097(93)90229-t. PMID 8459062
- [Background] Perez JE, Waggoner AD, Davila-Roman VG, Cardona H, Miller JG. On-line quantification of ventricular function during dobutamine stress echocardiography. Eur Heart J. 1992 Dec;13(12):1669-76. doi: 10.1093/oxfordjournals.eurheartj.a060123. PMID 1289098
- [Background] Rallidis L, Cokkinos P, Tousoulis D, Nihoyannopoulos P. Comparison of dobutamine and treadmill exercise echocardiography in inducing ischemia in patients with coronary artery disease. J Am Coll Cardiol. 1997 Dec;30(7):1660-8. doi: 10.1016/s0735-1097(97)00376-8. PMID 9385891
- [Background] Dagianti A, Penco M, Agati L, Sciomer S, Dagianti A, Rosanio S, Fedele F. Stress echocardiography: comparison of exercise, dipyridamole and dobutamine in detecting and predicting the extent of coronary artery disease. J Am Coll Cardiol. 1995 Jul;26(1):18-25. doi: 10.1016/0735-1097(95)00121-f. PMID 7797748
- [Background] Attenhofer CH, Pellikka PA, Oh JK, Roger VL, Sohn DW, Seward JB. Comparison of ischemic response during exercise and dobutamine echocardiography in patients with left main coronary artery disease. J Am Coll Cardiol. 1996 Apr;27(5):1171-7. doi: 10.1016/0735-1097(95)00583-8. PMID 8609338
- [Background] Olson CE, Porter TR, Deligonul U, Xie F, Anderson JR. Left ventricular volume changes during dobutamine stress echocardiography identify patients with more extensive coronary artery disease. J Am Coll Cardiol. 1994 Nov 1;24(5):1268-73. doi: 10.1016/0735-1097(94)90108-2. PMID 7930249
- [Background] Joseph T, Vieillard-Baron A, Chikli F, Goeau-Brissoniere O, Coggia M, Lacombe P, Dubourg O. Left ventricular volume analysis for the detection of coronary artery disease during dobutamine stress echocardiography in patients undergoing vascular surgery. Eur J Echocardiogr. 2000 Dec;1(4):263-70. doi: 10.1053/euje.2000.0039. PMID 11916604
- [Background] Coletta C, Galati A, Ricci R, Sestili A, Guagnozzi G, Re F, Ceci V. Prognostic value of left ventricular volume response during dobutamine stress echocardiography. Eur Heart J. 1997 Oct;18(10):1599-605. doi: 10.1093/oxfordjournals.eurheartj.a015139. PMID 9347270
- [Background] Rim SJ, Ha JW, Lee MH, Jang Y, Chung N. Left ventricular remodeling can be predicted with left ventricular volume response during dobutamine echocardiography after acute myocardial infarction. Clin Cardiol. 2008 Jun;31(6):259-64. doi: 10.1002/clc.20207. PMID 18543305
- [Background] Dagianti A, Rosanio S, Tocchi M, Trambaiolo P, Vitarelli A, Fedele F. [Left ventricular volumetric and contractility behavior during stress echocardiography with dobutamine]. Cardiologia. 1996 Mar;41(3):251-8. Italian. PMID 8697482
- [Background] Dehmer GJ, Lewis SE, Hillis LD, Corbett J, Parkey RW, Willerson JT. Exercise-induced alterations in left ventricular volumes and the pressure-volume relationship: a sensitive indicator of left ventricular dysfunction in patients with coronary artery disease. Circulation. 1981 May;63(5):1008-18. doi: 10.1161/01.cir.63.5.1008. No abstract available. PMID 7471358